CLINICAL TRIAL: NCT05800600
Title: Iron Replacement to Reduce Anemia During Neoadjuvant Chemotherapy
Acronym: Iron-RANC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-1053; HM-213 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venofer treatment (Experimental): Venofer (iron-sucrose) 200mg (5 days) every week administered as an IV infusion
  Interventions: Drug: Venofer

INTERVENTIONS:
Drug: Venofer — Intravenous iron will be administered as five doses of 200 mg of iron sucrose (Venofer, American Regent, Shirley, NJ) in 100 ml normal saline over a duration of 15 minutes to 1 hour

SUMMARY:
This is an open-label, single institution study evaluating the efficacy of intravenous iron sucrose monotherapy in patients with thoracic, breast, GU and GI malignancies undergoing neoadjuvant chemotherapy with the goal of undergoing surgical resection.

DETAILED DESCRIPTION:
This is an open-label, single institution study evaluating the efficacy of intravenous iron sucrose monotherapy in patients with thoracic, breast, GU and GI malignancies undergoing neoadjuvant chemotherapy with the goal of undergoing surgical resection. The concomitant use of radiation and immunotherapy as part of the neoadjuvant protocol is allowed in this protocol. The study is designed to evaluate the efficacy of iron infusions in reducing blood transfusion frequency and improving hemoglobin levels prior to surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years
* Patients undergoing neoadjuvant chemotherapy, including radiation and/or immunotherapy, with intent for curative surgical resection for breast, thoracic, gastrointestinal (GI) or genitourinary (GU) malignancies.
* Anemia defined as Hgb <10.5 g/dL during chemotherapy.
* Iron storage levels of ferritin <500 ng/mL and iron saturation <35%
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

* Diagnosis of anemia at the time of cycle 1 day 1 of neoadjuvant chemotherapy, Hgb < 11.0 g/dL, uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic new/exacerbated congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior parenteral iron infusion in the past 4 weeks
* The use of erythropoietin stimulating agents within 4 weeks unless chronic needs due to CKD
* Concurrent systemic infection at the time of enrollment.
* Known hypersensitivity to Iron sucrose
* Pregnant or breast feeding. Refer to section 4.4 for further detail.
* Anemia from another established etiology (i.e MDS, Myeloma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to highest Hgb value | 6 weeks
  To evaluate the efficacy of iron infusions in improving chemotherapy-induced anemia by improving the hemoglobin of patients undergoing neoadjuvant chemotherapy.
  Mean change from baseline to highest Hgb value observed six weeks after last iron infusion, before day of surgery.

SECONDARY OUTCOMES:
Number of transfusions during neo-adjuvant period | 24 weeks
  To evaluate the efficacy of iron infusions in improving chemotherapy-induced anemia and minimizing red blood cell transfusions in patients undergoing neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Iberia Sosa, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No